CLINICAL TRIAL: NCT05329909
Title: Epidemiology of Neurological Complications to Nitrous Oxide Poisoning
Acronym: EPI-NOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0023_NEURO; 2022-A00718-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-05

CONDITIONS: Neurology Department
Keywords: nitrous oxide poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
N2O inactivates vitamin B12, impairing its ability to act as a cofactor of methionine synthase. In addition, the elimination of vitamin B12 is increased. Neurological damage is similar to that described in combined sclerosis of the marrow, and are probably related to induce vitamin B12 deficiency. The use of N2O can then precipitate the rapid appearance of signs (neurological, psychiatric and hematological) related to a true and/ or functional vitamin B12 deficiency.

In 1978, RB Layzer described the first 3 cases of peripheral neuropathy secondary to nitrous oxide (N2O) consumption. In 2016, a team collected the 91 published cases: among these, 72 had neurological complications, and 52 had a concentration of vitamin B12 considered "low" or "normal-low"

Since then, consumption patterns seem changed due to: an increasing ease of access, the change of container (packaging in cartridge 8 grams versus bottle of 600 grams) and a usually occasional and festive consumption that seems to become solitary and regular, This change in consumption patterns is explained by an increased incidence of neurological complications, although no epidemiological work is yet available.

The objective of this work is to describe the epidemiology of this condition, to correlate it with major recent social phenomena (confinement related to the SARS-Cov2 pandemic), and finally to compare the incidence of myelopathies secondary to N2O with the incidence of other frequent inflammatory neurological diseases (autoimmune myelitis and Guillain-Barré syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥16 years)
* Hospitalized or having consulted with the departments of Neurology or Internal Medicine for neurological phenomena related to the consumption of N2O. The neurological phenomena included are usually: neuropathies or myelopathies, However, the existence of other neurological or psychiatric signs is not a factor of exclusion: for example, headaches or cognitive or psychiatric disorders with acute onset.
* Exposure to N2O for recreational or medical reasons (Meopa anesthesia).
* Lack of alternative diagnosis other than N2O poisoning
* Consultation for neurological disorders between 01/01/2018 and 31/12/2021

Exclusion Criteria:

* Minor subjects or subjects subject to a legal protection measure (guardianship, curators) during the consultation.
* Refusal to include in a study explained in the file
* Absence of N2O consumption during the 6 months preceding the appearance of signs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cohort of patients who have been exposed to N2O and have neurological disorders
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
sexe | Day 1
  describe the epidemiology of neurological complications to nitrous oxide poisoning
age | Day 1
  describe the epidemiology of neurological complications to nitrous oxide poisoning
place to live | Day 1
  describe the epidemiology of neurological complications to nitrous oxide poisoning
Occupational status | Day 1
  describe the epidemiology of neurological complications to nitrous oxide poisoning
consumption of toxic substances (alcohol, tobacco, cannabis) | Day 1
  describe the epidemiology of neurological complications to nitrous oxide poisoning

SECONDARY OUTCOMES:
Date and nature of first symptoms | Day 1
  correlate epidemiology with major recent social phenomena
consumption mode and quantity | Day 1
  correlate epidemiology with major recent social phenomena

OTHER OUTCOMES:
detail of symptoms, origin and consequences | Day 1
  compare the incidence of myelopathies secondary to N2O with the incidence of other frequent inflammatory neurological diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital DELAFONTAINE, Saint-Denis, Île-de-France Region, France

REFERENCES:
- [Background] Layzer RB, Fishman RA, Schafer JA. Neuropathy following abuse of nitrous oxide. Neurology. 1978 May;28(5):504-6. doi: 10.1212/wnl.28.5.504. PMID 205816
- [Background] Sanders RD, Weimann J, Maze M. Biologic effects of nitrous oxide: a mechanistic and toxicologic review. Anesthesiology. 2008 Oct;109(4):707-22. doi: 10.1097/ALN.0b013e3181870a17. PMID 18813051
- [Background] Garakani A, Jaffe RJ, Savla D, Welch AK, Protin CA, Bryson EO, McDowell DM. Neurologic, psychiatric, and other medical manifestations of nitrous oxide abuse: A systematic review of the case literature. Am J Addict. 2016 Aug;25(5):358-69. doi: 10.1111/ajad.12372. Epub 2016 Apr 1. PMID 27037733
- [Background] Vollhardt R, Mazoyer J, Bernardaud L, Haddad A, Jaubert P, Coman I, Manceau P, Mongin M, Degos B. Neurological consequences of recreational nitrous oxide abuse during SARS-CoV-2 pandemic. J Neurol. 2022 Apr;269(4):1921-1926. doi: 10.1007/s00415-021-10748-7. Epub 2021 Aug 21. PMID 34417869